CLINICAL TRIAL: NCT03719742
Title: A Clinical Study to Evaluate the Safety and Efficacy of a Baby Cleanser and a Moisturizer Under the Supervision of Dermatologist and Pediatrician
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of a Baby Cleanser and a Moisturizer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burt's Bees Inc. (Industry)
Collaborators: Stephens & Associates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: C18-D097
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sponsor Test Products (Experimental): 1. Baby Bee Foaming Cleanser(at least once daily)
  2. BB Baby Ultra Gentle Lotion (twice daily)
  Interventions: Other: Sponsor Test Products

INTERVENTIONS:
Other: Sponsor Test Products — Baby Bee Foaming Cleanser(at least once daily but not more than twice daily), BB Baby Ultra Gentle Lotion (Once immediately after cleansing and again approximately 10-12 hours after cleansing)

SUMMARY:
A Clinical Study to Evaluate the Safety and Efficacy of a Baby Cleanser and a Moisturizer Under the Supervision of Dermatologist and Pediatrician

DETAILED DESCRIPTION:
This single-center clinical trial is being conducted to demonstrate that the Sponsor's product does not statistically or clinically worsen eczema scores in children aged 6 months through 7 years after 4 weeks of treatment compared to baseline scores.

Safety and efficacy will be assessed through clinical grading at baseline and week 4. Efficacy will also be assessed through Corneometer and Tewameter measurements at baseline and week 4. Microbiome skin swab sampling will be performed at baseline and week 4. Parents/guardians will complete Patient Oriented Eczema Measure and Family Dermatology Quality of Life Index at baseline and week 4.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, female or male infants/children, aged 6 months through 7 years.
2. In generally good health (physical, mental, and social well-being, not merely the absence of disease/infirmity), according to parent/legal guardian report.
3. Having Fitzpatrick skin type I-VI (refer to Appendix I: Fitzpatrick Skin Type).
4. Having mild to moderate eczema involving 3% to 20% of body surface area, and with EASI score in the range of 1.1 to 20.0, further stratified into the following subgroups:

   * Approximately 60% of subjects with clinically determined EASI score of 1.1-7.0 (mild)
   * Approximately 40% of subjects with clinically determined EASI score of 7.1 to 20.0 (moderate)
5. Having a parent/legal guardian at least 18 years of age who regularly bathes the child and otherwise cares for the child, and who presents proof of guardianship (eg, insurance card, certificate of residence, or copy of officially issued family registration) at the baseline visit.
6. Having a parent/legal guardian willing to provide written informed consent and who can read, speak, write, and understand English.
7. Whose parent/legal guardian is willing to sign a photography release.
8. Willing, and having a parent/legal guardian who is willing, to cooperate and participate by following study requirements (including those outlined in section 7.3) for the duration of the study and to report any changes in health status or medications, AE symptoms, or reactions immediately.
9. Willing to bring in currently used moisturizer and cleanser to visit 1 for documentation by clinic staff.

Exclusion Criteria:

1. Diagnosed with known allergies to skin care products or ingredient(s) in the test product.
2. History of skin cancer within the past 5 years.
3. Individuals who have clinically active bacterial, fungal, or viral skin infections or those who have a history of recurrent cutaneous infections, according to subject self-report.
4. Individuals whose use of topical corticosteroids or systemic medications for their eczema has not been stable for at least 6 weeks prior to study start. This includes medicines such as hydrocortisone, clobetasol, betamethasone, halobetasol, fluocinide, diflorasone, mometasone, halcinonide, desoximetasone, pimecrolimus, tacrolimus, crisabarole, and fluticasone.
5. Having a health condition and/or pre-existing or dormant dermatologic disease on the body (eg, psoriasis, rosacea, acne [severe acne, acne conglobata, nodules, or cysts], seborrheic dermatitis, severe excoriations.) that the Investigator or designee deems inappropriate for participation or could interfere with the outcome of the study.
6. Who have observable suntan, scars, nevi, excessive hair, tattoos, or other dermal conditions on the body that might influence the test results in the opinion of the Investigator or designee.
7. Having a history of immunosuppression/immune deficiency disorders (including HIV infection, AIDS, multiple sclerosis, Crohn's disease, rheumatoid arthritis), had an organ transplant (heart, kidney, etc), or currently using oral or systemic immunosuppressive medications and biologics that are not used for the treatment of eczema (eg, azathioprine, belimumab, Cimzia, Cosentyx, cyclophosphamide, cyclosporine, Enbrel, Humira, Imuran, Kineret, mycophenolate mofetil, methotrexate, Orencia, Remicade, Rituxan, Siliq, Simponi, Stelara, Taltz) and/or undergoing radiation or chemotherapy as determined by study documentation.
8. Having a disease such as asthma, diabetes, epilepsy, hypertension, hyperthyroidism, or hypothyroidism that is not controlled by diet or medication; experiencing asthma flares or having multiple health conditions.
9. Having started a long-term medication within the last 2 months.
10. With any planned surgeries and/or invasive medical procedures during the course of the study. Non-invasive planned surgeries will be reviewed for their impact on the study outcome and acceptability by the Investigator or designee.
11. Who are currently participating in any other clinical trial at Stephens, another research facility, or doctor's office
12. Who have participated in any clinical trial or experimental treatment involving the test area within 4 weeks prior to inclusion into the study at Stephens, at another research facility or doctor's office.
13. Infants/children with a history of or exhibiting signs and symptoms of any systemic disease that may interfere with study evaluations (eg, urinary tract infections, significant bowel or urinary congenital malformation).
14. Infant/child who has had a recent change in her/his dietary intake or who has had severe diaper rash within 1 week prior to baseline.
15. Individuals who have received PUVA therapy for atopic dermatitis within 4 weeks prior to inclusion in the study.
16. Individuals who have received phototherapy within 2 weeks prior to inclusion in the study.
17. Individuals who have changed the type of moisturizer or cleanser used within the last 6 weeks prior to inclusion in the study.

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Eczema Area Severity Index (EASI) | 4 Weeks
  The primary efficacy endpoint is no worsening of the clinical appearance of atopic dermatitis/eczema as measured by the Eczema Area Severity Index (EASI) at week 4 from baseline. ranges from 0 (no eczema) to 72.

SECONDARY OUTCOMES:
The secondary endpoint is that the sponsors test materials will be well tolerated and well perceived by subject parents/guardians according to the Family Dermatology Quality of Life Index (FDQLI) | 4 Weeks
  Parent/Guardian Quality of Life as evaluated through subject parents/guardians according to the Family Dermatology Quality of Life Index (FDQLI). Scores range from 0-30. Measurement conducted at week 4 from baseline.

OTHER OUTCOMES:
No increase in transepidermal water loss values measured at Week 4 from baseline | 4 Weeks
  Transepidermal Water Loss. Tewameter measurements will be performed at baseline and week 4. A decrease in TEWL values reflects an improvement in the barrier properties of the skin.
No decrease in corneometry values at Week 4 from baseline | 4 Weeks
  Corneometer measurements will be performed at baseline and week 4. The measurement has no units, but is proportional to the dielectric constant of the surface layers of the skin, and increases as the skin becomes more hydrated.

CONTACTS AND LOCATIONS:
Overall Officials: Lily Jiang, PhD, Principal Investigator — Stephens & Associates, Inc.
Locations (1):
- Stephens & Associates, Inc, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No